CLINICAL TRIAL: NCT04587167
Title: HPV ECHO: Increasing the Adoption of Evidence-based Communication Strategies for HPV Vaccination in Rural Primary Care Practices
Brief Title: HPV Vaccine Communication ECHO for Primary Care Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, William Calo, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00015734; R37CA253279 (NIH)
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Human Papillomavirus Vaccines; Adolescent Health Services

STUDY DESIGN:
Intervention Model Description: Cluster randomized design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HPV ECHO (Experimental): Clinics randomly assigned to this arm will receive the intervention via real-time, interactive videoconferencing using Zoom at no cost to participants. The intervention has a curriculum of 10 sessions focused on the evidence-based Announcement Approach. Sessions will be 60 minutes in duration and held every other weekly for 4 months at regularly scheduled times.
  Interventions: Other: Project ECHO; Other: Announcement Approach Training
- HPV ECHO+ (Experimental): Clinics randomly assigned to this arm will receive the HPV ECHO intervention plus a systems communication strategy to deliver recall notices to parents who initially decline HPV vaccination. This arm includes 12 primary care clinics in Pennsylvania.
  Interventions: Other: Project ECHO; Other: Announcement Approach Training; Other: Recall notices
- Control (No Intervention): Clinics randomly assigned to this arm will receive no ECHO interventions. This arm includes 12 primary care clinics in Pennsylvania.

INTERVENTIONS:
Other: Project ECHO — Using proven adult learning techniques and interactive video technology, the ECHO Model promotes knowledge exchange between experts or specialists at centers of excellence ("the hub") and primary care providers (the "spokes), typically located in rural settings. Through regular real-time collaborative sessions, the spokes connect with the hub and with other spokes to discuss 1) best practices in care and 2) complex cases managed within their practice.
  Other Names: ECHO Model
  Arms: HPV ECHO; HPV ECHO+
Other: Announcement Approach Training — Train physicians and their clinic staff to make strong HPV vaccine recommendations by using presumptive announcements. If parents show vaccine hesitancy, the Training train physicians a 3-step approach (Connect, Clarify, Counsel) to share effective, evidence-based messages about HPV vaccine.
  Arms: HPV ECHO; HPV ECHO+
Other: Recall notices — Notify parents that their child is behind for HPV vaccination. Recall notices will include research-tested messages to specifically address parent concerns. Recall notices will be sent to parents via patient portal or email communication.
  Arms: HPV ECHO+

SUMMARY:
The safe, highly-effective human papillomavirus (HPV) vaccine remains underused in the US; only 51% of 13- to 17-year-old girls and boys were up-to-date by 2018. The Announcement Approach Training is effective in increasing HPV vaccine uptake during the clinic visit by training providers to make strong vaccine recommendations and answer parents' common questions. Systems communication like recall notifications also improve vaccination by reducing missed clinical opportunities. Although never tested to support HPV vaccination, the ECHO (Extension for Community Healthcare Outcomes) Model is a proven implementation strategy to promote capacity exchange between health care experts at academic centers and primary care providers at the front line of rural community health care. The trial will test the effectiveness of two ECHO-delivered HPV vaccination communication interventions versus control: HPV ECHO will provide Announcement Approach training, and HPV ECHO+ will provide training plus recall notices to communicate with parents who initially decline vaccination.

DETAILED DESCRIPTION:
The investigators will recruit 36 primary care clinics (family medicine and pediatric) in Pennsylvania. Eligible clinics will have at least 100 active patients, ages 11-14, in their electronic health record systems. Recruitment will target clinics in Central Pennsylvania, where most counties are designated as rural. Clinics will be randomized to one of three arms: ECHO-delivered HPV vaccine communication training using the Announcement Approach (HPV ECHO); HPV ECHO plus systems follow-up communication for parents who initially decline vaccination (HPV ECHO+); or control. Covariate-constrained randomization will be used to ensure balance among the three arms with respect to clinic size (adolescent patient population), clinic type (academic vs. non-academic), rurality, and historic adolescent HPV vaccination rates.

ELIGIBILITY:
Clinics in cluster RCT (main study)

Inclusion Criteria:

* Family medicine or pediatric clinic in Pennsylvania
* Having at least 100 active patients, ages 11-14.

Exclusion Criteria:

* Primary care clinic outside Pennsylvania
* Participated in HPV vaccine communication or quality improvement research either through Penn State or another institution in the last 12 months.

Parents in nested study survey

Inclusion criteria:

* Parent or guardian of an adolescent ages 11-17
* Adolescent has not yet started HPV vaccination
* Adolescent receive primary care at participating clinic

Exclusion criteria:

* Not the parent or guardian of an adolescent ages 11-17
* Adolescent already initiated HPV vaccination
* Adolescent does not receive primary care at participating clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
HPV vaccination (≥1 dose), 11-14 year olds at 12 months | Twelve months
  Coverage change from baseline to 12 months in HPV vaccine initiation (≥1 dose), among 11- to 14- year old patients, as measured by clinics' records

SECONDARY OUTCOMES:
HPV vaccination (≥1 dose), 11-14 year olds at 3 months | Three months
  Coverage change from baseline to 3 months in HPV vaccine initiation (≥1 dose), among 11- to 14- year old patients, as measured by clinics' records
HPV vaccination (≥1 dose), 11-14 year olds at 6 months | Six months
  Coverage change from baseline to 6 months in HPV vaccine initiation (≥1 dose), among 11- to 14- year old patients, as measured by clinics' records
HPV vaccination (≥1 dose), 11-14 year olds at 9 months | Nine months
  Coverage change from baseline to 9 months in HPV vaccine initiation (≥1 dose), among 11- to 14- year old patients, as measured by clinics' records
HPV vaccination (completion), 11-14 year olds at 3 months | Three months
  Coverage change from baseline to 3 months in HPV vaccine completion (according to the Advisory Committee on Immunization Practices (ACIP) guidelines), among 11- to 14- year-old patients, as measured by clinics' records
HPV vaccination (completion), 11-14 year olds at 6 months | Six months
  Coverage change from baseline to 6 months in HPV vaccine completion (according to the Advisory Committee on Immunization Practices (ACIP) guidelines), among 11- to 14- year-old patients, as measured by clinics' records
HPV vaccination (completion), 11-14 year olds at 9 months | Nine months
  Coverage change from baseline to 9 months in HPV vaccine completion (according to the Advisory Committee on Immunization Practices (ACIP) guidelines), among 11- to 14- year-old patients, as measured by clinics' records
HPV vaccination (completion), 11-14 year olds at 12 months | Twelve months
  Coverage change from baseline to 12 months in HPV vaccine completion (according to the Advisory Committee on Immunization Practices (ACIP) guidelines), among 11- to 14- year-old patients, as measured by clinics' records
HPV vaccination (≥1 dose), 15-17 year olds at 3 months | Three months
  Coverage change from baseline to 3 months in HPV vaccine initiation (≥1 dose), among 15- to 17- year old patients, as measured by clinics' records
HPV vaccination (≥1 dose), 15-17 year olds at 6 months | Six months
  Coverage change from baseline to 6 months in HPV vaccine initiation (≥1 dose), among 15- to 17- year old patients, as measured by clinics' records
HPV vaccination (≥1 dose), 15-17 year olds at 9 months | Nine months
  Coverage change from baseline to 9 months in HPV vaccine initiation (≥1 dose), among 15- to 17- year old patients, as measured by clinics' records
HPV vaccination (≥1 dose), 15-17 year olds at 12 months | Twelve months
  Coverage change from baseline to 12 months in HPV vaccine initiation (≥1 dose), among 15- to 17- year old patients, as measured by clinics' records
HPV vaccination (≥1 dose), 11-14 year olds at 12 months by sex | Twelve months
  Coverage change from baseline to 12 months in HPV vaccine initiation (≥1 dose), among 11- to 14- year old patients by sex, as measured by clinics' records
HPV vaccination (≥1 dose), 15-17 year olds at 12 months by sex | Twelve months
  Coverage change from baseline to 12 months in HPV vaccine initiation (≥1 dose), among 15- to 17- year old patients by sex, as measured by clinics' records

OTHER OUTCOMES:
Tetanus, diphtheria, and acellular pertussis (Tdap) vaccination, 11-14 year olds | Twelve months
  Coverage change from baseline to 12 months in Tdap vaccination among 11- to 14-year-old patients, as measured by clinics' records
Meningococcal vaccination (≥1 dose), 11-14 year olds | Twelve months
  Coverage change from baseline to 12 months in meningococcal vaccination (≥1 dose), among 11- to 14-year-old patients, as measured by clinics' records

CONTACTS AND LOCATIONS:
Overall Officials: William A Calo, PhD, JD, MPH, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No raw data will be shared with the general public or other researchers.

REFERENCES:
- [Derived] Calo WA, Shah PD, Fogel BN, Ruffin Iv MT, Moss JL, Hausman BL, Segel JE, Francis E, Schaefer E, Bufalini CM, Johnston N, Hogentogler E, Kraschnewski JL. Increasing the adoption of evidence-based communication practices for HPV vaccination in primary care clinics: The HPV ECHO study protocol for a cluster randomized controlled trial. Contemp Clin Trials. 2023 Aug;131:107266. doi: 10.1016/j.cct.2023.107266. Epub 2023 Jun 9. PMID 37301468